CLINICAL TRIAL: NCT01295593
Title: Phase I-II Study of Low Dose CdA Combined With Valproic Acid (VPA) in Previously Treated B-cell Chronic Lymphocytic Leukemia (CLL) Patients
Brief Title: Low Dose CdA Combined With Valproic Acid (VPA) in Previously Treated B-cell Chronic Lymphocytic Leukemia(B-CLL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPA-CdA
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL previously treated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Valproic Acid; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valproic acid combined with CdA (Experimental): valproic acid, oral daily intake, combined with 2-chlorodeoxyadenosine administered intravenously for 4 cycles
  Interventions: Drug: valproic acid and 2-chlorodeoxyadenosine

INTERVENTIONS:
Drug: valproic acid and 2-chlorodeoxyadenosine — VPA : daily, oral, starting dose 10mg/kg/day total dose, taken in 2 separate administrations of around 5 mg/kg/day each, for a maximum of 6 months CdA : 5.6 mg/m²/day IV during 3 days, every 28 days, for a maximum of 4 cycles

SUMMARY:
Rationale New chemotherapeutic agents are needed in relapsing B-Cell Chronic Lymphocytic Leukemia (B-CLL) to overcome resistance of CLL cells. Valproic acid (VPA) is an inhibitor of histone deacetylase (HDAC) used as an anticonvulsant and mood-stabilizing drug for decades. VPA mediates apoptosis in CLL cells through caspase activation. VPA shows toxicity toward CLL cells displaying alterations in the p53 pathway. The combination of VPA with fludarabine or 2-Chlorodeoxyadenosine (CdA, Cladribine) results in synergistic loss of B-CLL cell viability, and significant increase in apoptosis. The highest index of synergism is observed between VPA and CdA, a purine nucleoside analog active in B-CLL.

Study design Overall, the study will be proposed to previously treated patients with advanced B-CLL, who are not eligible for aggressive approaches, and who exhibit progressive disease. A total of 33 patients will be included. Estimated enrolment time is 2 years.

* First part: It is planned to start therapy with single VPA during 2 months, targeting plasma levels that have been reported to be active in vitro toward CLL cells (but that do not exceed therapeutic levels in seizure prevention), and in parallel, to verify whether cellular targets of VPA have been actually inhibited in leukemic B-lymphocytes.
* Second part: After the VPA preloading period (2 months), patients will be evaluated to receive CdA. CdA will be given at 5.6 mg/m²/day intravenously during 3 days, a reduced-dose schedule which is less toxic - at no obvious cost of loss of efficacy - as compared to the standard dosage of 5 days. CdA was chosen because it displays the highest level of in vitro synergism with VPA. Four monthly courses of CdA will be given. Patients will then be evaluated. VPA will be stopped at the time of response evaluation (scheduled 28 days after the last course of CdA).

ELIGIBILITY:
Inclusion Criteria:

* B-cell Chronic Lymphocytic Leukemia (CLL)
* Patients must have intermediate or high-risk categories of the modified 3-stage Rai and Binet staging
* Patient MUST have progressive or symptomatic disease as defined by any of the following conditions:

  * Progressive lymphocytosis with a lymphocyte count increased > 50% over the last 2 months period or an anticipation of the doubling time in less than 6 months
  * Progressive or symptomatic splenomegaly or hepatomegaly
  * Progressive or symptomatic lymphadenopathy
  * Evidence of progressive marrow failure as manifested by development or worsening of anemia and/or thrombocytopenia
  * Presence of any B-symptoms: weight loss ≥ 10% within the previous 6 months, fever > 38.0°C for ≥ 2 weeks without evidence of infection, or night sweats without evidence of infection
* Patient must have received one or more prior therapies for Chronic Lymphocytic Leukemia. Patients may have received any of the following prior treatment regimens: fludarabine-containing combinations, alemtuzumab single agent or combination, rituximab combinations, chlorambucil, cyclophosphamide +/- prednisone, or other forms of immunotherapy…
* Patients must have adequate organ function:

  * Neutrophils > 500/mm³
  * Platelets > 50.000/mm³
  * Creatinine clearance (measured or calculated) > 40 ml/min
* Age > 18 years
* Patient's ECOG performance status must be 0-2
* Patient's written informed consent
* Life expectancy > 6 months

Exclusion Criteria:

* Patients having received Valproic Acid (VPA) within 3 months
* Previous, suspected or known hypersensitivity to VPA, or any of its derivatives
* Liver porphyria
* Epilepsy due to mitochondrial diseases
* Ongoing treatment with VPA-interacting drugs
* Cumulative Illness rating Scale (CIRS) > 6
* Prior allogenic or autologous bone marrow transplantation less than 12 months
* Patient having received any anticancer agents (chemotherapy, immunotherapy or targeted agents) within 4 weeks
* Central Nervous System involvement
* Concomitant disease requiring prolonged use of corticosteroids (> 1 month)
* Transformation into an aggressive B-cell malignancy (e.g. diffuse large cell lymphoma, Hodgkin lymphoma)
* Creatinine clearance < 40 ml/min calculated according to the formula of Cockcroft and Gault. Patients with a calculated creatinine clearance below 40 ml/min may be eligible if (1) a measured creatinine clearance (based on 24 hours urine collection or other reliable method) is > 40 ml/min, or (2) a new calculation conducted after adequate hydration is > 40 ml/min.
* Any coexisting medical or psychological condition that would preclude participation to the required study procedures
* Patient with mental deficiency preventing proper understanding of the requirements of treatment
* Pregnancy, lactating woman, females of childbearing potential or male patient who are unwilling to use adequate contraception
* Clinically significant auto-immune cytopenia, Coombs-positive hemolytic anemia as judged by the treating physician
* Patients with a history of another malignancy in complete remission less than 2 years, except basal cell skin cancer, stage 0 (in situ) cervical carcinoma or tumor treated curatively by surgery
* Any severe co-morbidities such as New York Heart Association Class III or IV heart failure, myocardial infarction within 6 months, unstable angina, ventricular tachyarrhythmias requiring ongoing treatment, or severe uncontrolled myocardiopathy, uncontrolled hypertension, severe chronic obstructive pulmonary disease with hypoxemia or uncontrolled diabetes mellitus
* Active bacterial, viral or fungal infection
* Seropositivity for: Human Immunodeficiency Virus, hepatitis C or hepatitis B (unless clearly due to vaccination)
* Liver insufficiency
* Total bilirubin > 2 x the upper limit of normal (ULN)
* Prior history of severe hepatic or pancreatic disorder
* Alkaline phosphatases and aminotransferases (AST, ALT) > 2 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
To determine the tolerability of VPA in combination with low dose CdA in patients with advanced B-CLL | 6 months on average

SECONDARY OUTCOMES:
minimal dose of VPA able to achieve adequate plasma levels of VPA and effective inhibition of VPA cellular targets, therapeutic response and survival , VPA pharmacokinetics | 6 months on average

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Den Neste, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (11):
- Belgium (11):
  - Clinique Sud Luxembourg, Arlon
  - Institut Jules Bordet, Brussels
  - ULB Erasme, Brussels
  - Cliniques universitaires Saint Luc, Brussels
  - Grand Hôpital de Charleori - Site notre Dame, Charleroi
  - Clinique Notre-Dame de Grâce, Gosselies
  - Hôpital de Jolimont, Haine-St-Paul
  - CHU ULg, Liège
  - Clinique Saint Pierre, Ottignies
  - Heilig-Hartziekenhuis, Roeselaere
  - Cliniques de Mont Godinne, Yvoir